CLINICAL TRIAL: NCT00093769
Title: A Phase II Study of VELCADE With Rituximab in Subjects With Relapsed or Refractory Indolent B-Cell Lymphoma
Brief Title: Bortezomib and Rituximab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000390235; UCLA-0401054-01; MILLENNIUM-M34103-061
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib; Rituximab

ARMS (1):
- bortezomib + rituximab (Experimental): Arm I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Patients also receive rituximab IV on days 1, 8, and 15 of course 1 only and on day 1 of course 2 only. Treatment with repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Arm II: Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15 and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 only. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients in either arm may crossover to the other arm if treatment is found to be ineffective.
  Interventions: Drug: bortezomib + rituximab

INTERVENTIONS:
Drug: bortezomib + rituximab — Arm I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Patients also receive rituximab IV on days 1, 8, and 15 of course 1 only and on day 1 of course 2 only. Treatment with repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15 and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 only. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Patients in either arm may crossover to the other arm if treatment is found to be ineffective.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Giving bortezomib together with rituximab may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying how well giving bortezomib together with rituximab works in treating patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete response [CR], CR-unconfirmed [CRu], and partial response [PR]) in patients with relapsed or refractory indolent B-cell non-Hodgkin's lymphoma treated with bortezomib and rituximab.

Secondary

* Determine the response rate (CR, CRu, and PR) at the first disease response evaluation in patients treated with this regimen.
* Determine the overall CR rate (CR and CRu) in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the time to best response in patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, Karnofsky performance status (< 70% vs ≥ 70%), lactic dehydrogenase level (normal vs > upper limit of normal), age (18 to 60 years vs > 60 years), and lymphoma subtype (follicular vs marginal zone). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Patients also receive rituximab IV on days 1, 8, and 15 of course 1 only and on day 1 of course 2 only. Treatment with repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15 and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 only. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients in either arm may crossover to the other arm if treatment is found to be ineffective.

Patients are followed at 30 days and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 24-66 patients (12-33 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of indolent B-cell non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Follicular (grade 1, 2, or 3)
  * Marginal zone (extranodal, nodal, or splenic)
* CD20-positive disease
* Relapsed or progressive disease after prior anti-neoplastic therapy, as indicated by 1 of the following:

  * New lesions
  * Objective evidence of progression of existing lesions
* Complete response ≥ 6 months in duration after prior rituximab therapy* NOTE: *For patients who were previously treated with a regimen that included rituximab
* At least 1 measurable lymph node mass > 1.5 cm in 2 perpendicular dimensions that has not been irradiated OR that has progressed since prior radiotherapy
* No active CNS lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 50-100% OR
* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 50,000/mm^3

Hepatic

* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN

Renal

* Creatinine ≤ 2 mg/dL OR
* Creatinine clearance ≥ 30 mL/min

Immunologic

* No known anaphylaxis or immunoglobulin E-mediated hypersensitivity to murine proteins or to any component of rituximab, including polysorbate 80 and sodium citrate dihydrate
* No active systemic infection requiring treatment
* No history of allergic reaction attributable to compounds containing boron or mannitol

Other

* No peripheral neuropathy or neuropathic pain ≥ grade 2
* No other malignancy within the past 5 years except completely resected basal cell or squamous cell skin cancer or an in situ malignancy

  * Previously diagnosed prostate cancer allowed provided the following criteria are met:

    * T1-2a, N0, M0 disease AND Gleason score ≤ 7 AND prostate specific antigen (PSA) ≤ 10 ng/mL before initial therapy
    * Treated with definitive curative therapy (i.e., prostatectomy or radiotherapy) within the past 2 years
    * No clinical evidence of prostate cancer AND undetectable PSA (for prostatectomy patients) or PSA < 1 ng/mL (for patients who did not undergo prostatectomy)
* No serious medical or psychiatric illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 10 weeks since prior radioimmunoconjugates or toxin immunoconjugates (e.g., ibritumomab tiuxetan or iodine I 131 tositumomab)
* More than 4 weeks since prior rituximab, alemtuzumab, or other unconjugated therapeutic antibody
* No concurrent prophylactic bone marrow growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or epoetin alfa) during course 1 of study therapy

Chemotherapy

* More than 6 weeks since prior nitrosoureas
* No concurrent cisplatin

Endocrine therapy

* No concurrent corticosteroids (e.g., dexamethasone) except prednisone ≤ 15 mg/day or equivalent for adrenal insufficiency

Radiotherapy

* See Disease Characteristics
* See Biologic therapy
* More than 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 2 weeks since prior major surgery

Other

* Recovered from all prior therapy
* No prior bortezomib
* More than 3 weeks since prior antineoplastic therapy
* More than 3 weeks since prior experimental therapy
* No other concurrent antineoplastic therapy
* No other concurrent investigational agents

  * Concurrent participation in a non-treatment study allowed provided it does not interfere with participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response [CR], CR-unconfirmed [CRu], and partial response [PR]) | 12 weeks

SECONDARY OUTCOMES:
Response rate (CR, CRu, and PR) at the first disease response evaluation | 12 weeks
Overall CR rate (CR and CRu) | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sven De Vos, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] de Vos S, Goy A, Dakhil SR, Saleh MN, McLaughlin P, Belt R, Flowers CR, Knapp M, Hart L, Patel-Donnelly D, Glenn M, Gregory SA, Holladay C, Zhang T, Boral AL. Multicenter randomized phase II study of weekly or twice-weekly bortezomib plus rituximab in patients with relapsed or refractory follicular or marginal-zone B-cell lymphoma. J Clin Oncol. 2009 Oct 20;27(30):5023-30. doi: 10.1200/JCO.2008.17.7980. Epub 2009 Sep 21. PMID 19770386